CLINICAL TRIAL: NCT04884711
Title: Designing New Dignified Technologies for Care Settings in Participation With Older People.
Brief Title: INNOVATEDIGNITY: Co-designing Digital Health Technologies With Older People in Homecare Settings.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Brighton (Other)
Collaborators: Brighton & Hove Digital Health Living Lab (Unknown); Nord University (Other)
Responsible Party: Principal Investigator, Prof. Kathleen Galvin, Professor of Nursing Practice, University of Brighton
Other Study IDs: 2020-5669; 813928 (Other Grant/Funding Number: European Commission)
Record Dates: First submitted 2020-11-20; First posted 2021-05-13 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Dignity; Old Age; Debility; Healthy Aging; Digital Technology
Keywords: geriatrics; wearable electronic devices; self-help devices; biomedical technology; disruptive technology; Healthy Ageing; aged; homes for the aged; Human Centered Design; Digital Technology
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Interviews: Older people living at the Leach Court (Brighton, UK).: Older adults who will be enrolled at the Leach Court (Brighton, UK) as a part of the INNOVATEDIGNITY project will be involved in 1:1 open ended interviews.
  Interventions: Other: No Interventions. Participants will be using their everyday digital health technologies.; Other: In depth Interviews
- Focus Group Discussions: Older People Living at the Leach Court (Brighton, UK): 10 older people who have previously participated in the interview stage will be involved in two focus group discussions in a group of 5 participants each to co-design digital health technologies that are 'dignity' sensitive and aims to resolve the barriers older people face in technology adoption.
  Interventions: Other: Focus Group Discussions

INTERVENTIONS:
Other: No Interventions. Participants will be using their everyday digital health technologies. — The investigators will be involving older people to understand the barriers & facilitators of digital health technology adoption for homebound older people. In this process no interventions will be given by us.
  Groups: Interviews: Older people living at the Leach Court (Brighton, UK).
Other: In depth Interviews — In-depth interviews will be conducted to gather lived experiences of homebound older people.
  Groups: Interviews: Older people living at the Leach Court (Brighton, UK).
Other: Focus Group Discussions — Focus Group Discussions will be used to create avenues to enhance dignity and human perspectives in digital designs for older people.
  Groups: Focus Group Discussions: Older People Living at the Leach Court (Brighton, UK)

SUMMARY:
One of the crucial components of successful ageing is to live independently in old age. Yet in UK alone, nearly 300000 older people require assistance with 3 or more essential daily tasks like eating, bathing and mobility which compromises on their independent living. Additionally, in a crisis where health system in UK is already overstretched to its resources to combat the recent Coronavirus Disease 2019 (COVID-19) pandemic, allocating resources for regular homecare services has become challenging. In this situation, Digital Health Technologies (DHTs) can be a potential solution to promote healthy ageing, support psycho-social wellbeing and enhance independent living for older people. Such technologies comprise a wide range of products used in the health and care services including apps, software and online platforms to benefit people. Yet DHTs are barely adopted by older people as they do not reflect their actual user needs leading to poor appropriation of DHTs in homecare settings. The investigators aim to address this gap by involving older people living at the Leach Court, UK under the eco system of the Brighton & Hove Digital Health Living Lab (BHLL) to co-design with us DHTs that addresses the barriers & facilitators they face in adopting to DHTs. This participatory research approach has a qualitative study design which is sensitive to basic human values like 'dignity', appreciates that older people are 'expert of their experiences' and methodologically has phenomenological underpinnings gathering the researcher's understanding from the lived experiences of older people. This unique project, part of the European Union (EU) Horizon 2020 funded INNOVATEDIGNITY project, will be aiming to translate intangible human values like 'dignity' into tangible technology design through better understanding of the barriers & facilitators older people face to DHTs adoption. With global population of older people increasing faster than all other age groups currently, this project stands to meet the future demands of the ageing population through dignity sensitive better designed DHTs .

This project is part of the Marie Skłodowska-Curie Actions (MSCA) Innovative Training Networks (ITN). This project has received funding from the European Union's H2020-MSCA-ITN-2018 programme under grant agreement No 813928.

DETAILED DESCRIPTION:
Background:

Older people (65 years & above) in UK comprised of 17.8% of the total population (11.3 million) in 2014 with nearly 300000 older people within this group requiring help with 3 or more essential daily tasks. With progressive age older people are increasingly preferring to age in place as in home care settings with possibilities of higher dependence on digital health technologies . Yet such technologies are barely adopted by older people as they do not reflect actual user needs. The inappropriateness of these products at many times compromises on human dignity leading to poor adoption.

Designing digital health technologies for the older people living in care settings present significant challenges in terms of defining such technologies in the design process, establishing their needs in the relevant care settings and recruiting appropriate group of study participants. In fact, evidence points towards studies where care providers, family members, physicians and technologists were key participants which failed to portray the actual needs of older people. Worst still, technology design studies are mostly conducted in corporate showrooms or simulated research laboratories which are inadequate to capture real life settings. Therefore, there is a need for studies that involves older people to create acceptable, adoptable & adaptable digital health technologies for them.

Furthermore, designing such products for older people also presents challenges in terms of data privacy, training necessities for upgraded products, complex user interfaces and faulty devices malfunctioning under complex situations. In a qualitative study engaging older people of Finland and Spain to explore ethical and privacy related issues around 3 instrumental activities of daily living (monitoring the taking of medication, sleep monitoring & home security) found respondents concerned about product costs, data privacy, data confidentiality and possibilities of their autonomy being challenged. Moreover, respondents raised questions about devices giving false notifications and alarms.

The above stated issues show that there is a significant need to rethink design considerations of dignified technologies for older people mainly because actual perceptions of older people are not taken into design considerations leading to poor technology uptake. From broader perspectives, it can potentially reduce workload of healthcare professionals, improve data collection from care settings, enhance communication across levels of care and optimize health expenditure for UK. Therefore, there is a significant importance & possibility to address the present research gap by including the actual perceptions of older people in the design process and create technology infused with human factors & dignity to promote their independent living.

Research Aim:

To co-design new dignified technologies for care settings in participation with older people living in the Leach Court, Brighton which is part of the open innovation ecosystem of the Brighton & Hove Digital Health Living Lab(BHLL), an enterprise project of the University of Brighton.

Specific Objectives:

1. To appraise the existing scientific evidence on using participatory approach to create digital health technologies for older people in care settings.
2. To explore the perceptions of older people on using digital health technologies for activities of daily needs.
3. To analyze the facilitators & barriers of digital health technology uptake for older people living in care settings.
4. To identify strategies to enhance dignity and human perspectives in digital design for older people living in care settings.
5. To recommend relevant outcomes of the study to stakeholders for implementation in UK.

Research Design:

The present qualitative study uses phenomenologically led participatory design approach to involve older people (participants) living in a supported housing facility at the Leach Court (Brighton, UK) to understand from their lived experiences the barriers & facilitators they face in digital health technology adoption in everyday life and further, consider them to use their experience to conceptually co-design with the research team future dignified digital health technologies that fulfills their needs.

Research Methods:

1. Eligibility Assessment: - A participant questionnaire will be used to screen candidates for the study based on the eligibility criteria. However, the research team will also consider older people with no exposure to digital health technologies as that can offer considerable insight on the barriers to digital health technology adoption for older people.
2. Face to Face Interviews: 1:1 qualitative open ended interviews will be conducted preferably at the residence of the participants using phenomenologically led reflective lifeworld approach. About 2 weeks prior to the interview, participants will be provided with a 'prompt resource pack' containing an instant analog camera which will be used by participants to capture photos of digital health technologies they use in everyday life. Photographs can evoke deeper experiences revealing the latent & tacit needs of the users. Thereby, strengthening the data collection for this study through a photovoice approach.

   These pictures will be used as probing tools during the interview sessions to gather rich data to identify the barriers and facilitators of technology adoption for older people. Participants will be observed & documented for their non-verbal communication during the interview. Participants may be approached for subsequent interviews to reveal better understanding of the phenomenon of digital health technology adoption.
3. Co-design Workshops: 1 month prior to the co-design workshops the investigators will conduct an awareness seminar which will aim at sensitizing older people about diverse types of digital health technologies. Purpose of such a seminar will be to raise the consciousness of participants on such technologies. In Co-design workshops, qualitative focus group discussions (FGD) based on underpinnings of dialogal phenomenology will be held with older people who have been part of the earlier data collection process of this study. The purpose will be to create strategies that can improve acceptance and address dignity issues with digital health technologies for older people.

COVID-19 Contingency Plan for Data Collection:

In case there is uncertainty in collecting data through face to face interviews and other methods as has been outlined earlier, the research team will collect data through University of Brighton's approved online data gathering approaches. This is a forecast based on the present COVID-19 pandemic situation across the globe.

Data Analysis:

Anonymised data will be analysed phenomenologically to reveal core and unique aspects of the phenomenon under study. Data from interviews will be analyzed using principles of 'reflective lifeworld approach' whereby anonymised data will be read multiple times to gain data familiarity. The text will be subdivided into segments of meaningful units. While reading the text the site-investigator will be moving back & forth within the data to organize parts of the whole text in order to see patterns that describe the phenomenon in a logical way to reveal core & unique aspects of the phenomenon. This is termed as 'whole-parts-whole' approach.

Data from Co-Design workshop will be analysed using principles of dialogal phenomenology.

Ethical Considerations:

The study has been approved a favorable ethical opinion based on the details provided above from the Life,Health & Physical Sciences College Research Ethics Committee (CREC) of University of Brighton (UK). For consideration of ethical issues pertaining to the project the investigators have considered the possible vulnerabilities of older people on the ethical principles of autonomy, beneficence, non-maleficence and justice. The investigators will perform capacity interviewing at appropriate points during data collection process to ascertain the participant's capacity to consent for the study. Participant Information Sheets (PIS) will be provided before all data collection steps so that participants are aware of the objectives, purpose and process of the study. Informed Consent will be sought after explaining the PIS to participants and attending to any query from participants that may be relevant to the study. Participation will be completely voluntary and participants can resign from the study at any point without citing any reasons. Only anonymised data will be analyzed and confidentiality of participants will be retained.

Previous Clinical Trials:

In the context of this study, the clinical trials database was searched to ascertain that this study was not a duplication of previous studies. The search of clinical trials database revealed few studies exploring lived experiences, working on digital health interventions and co-designing of technologies but none were concerned with dignity perspectives in relation to digital health technologies. All such trials are provided with an unique National Clinical Trial (NCT) number.

In terms of lived experiences, two studies were concerned with children (NCT00456209 & NCT04168515). Most were concerned with health conditions & diseases like Irritable Bowel Disease (IBD), mental health, prostate cancer etc. (NCT04274725,NCT03131505, NCT02889536,NCT04399096 & NCT02690272). Few were focused on lived experiences of health professionals (NCT04168515 & NCT03709537). One study was primarily focused on lived experiences of older people but did not constitute dignity perspectives in digital health technology adoption (NCT04503811). One study was identified with co-learning approach for mental health workforce but this was not related to aged people (NCT03709537).

In terms of digital health, two studies related to the domain of co-designing could be identified. One involved older people to create a 'digital bridge' (NCT04287192) and another focused on involving care professionals to improve transitions from stroke unit to the home (NCT02925871). Another study could be located which involved older people in Accident & Emergency Department in a hospital but not in homecare settings (NCT04085796).

The investigators could locate one clinical trial on studying the perception changes of personal dignity during progression of dementia in patients but that study was not involved with any digital health technologies (NCT04443621).

The review of the existing evidence base on clinical trials reveal that this study is unique in involving homebound older adults in a co-design approach to improve digital health technology adoption and enhancing dignity perspectives in digital design.

Funding Information:

This project has received funding from the European Union's H2020-MSCA-ITN-2018 programme under grant agreement No 813928.

ELIGIBILITY:
Inclusion Criteria:

* Age should be at least 65 years.
* Participants who are able to read & write in English.
* Older people living in the Leach Court (Brighton, UK) for at least the past one year.
* Participants of all gender will be entertained.

Exclusion Criteria:

* People who are unable to communicate in english.
* Older People with terminal illness and profound cognitive disabilities will be excluded as their inclusion might be challenged by age related frailty, poor communication and life threatening medical conditions. However, benefits of the research will be extended to them by sharing the research outcomes.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — The investigators will welcome an inclusive approach to technology design by involving people from all gender based on their self-identification.
Study Population: Older adults meeting the inclusion criteria and living in the Leach Court (Brighton, UK). There will be 10 older participants in this study and if many more people volunteers, the investigators will invite a maximum of 20 participants.
  Participants will be selected based on age range, gender, existing disabilities, and exposure to digital health technologies. The research plans for at least 2 participants per chronologically advancing age group inter spaced at a 5 years interval starting from 65- 70 years & ending at 85-90 years. The participants will be gradually recruited as responses arrive with the research investigator. The study group is vulnerable especially in the light of current COVID 19 crisis with multiple underlying co-morbid conditions.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2021-07-30 (Estimated); Primary Completion 2021-09-15 (Estimated); Study Completion 2021-09-15 (Estimated)

PRIMARY OUTCOMES:
Participants Lived Experience with Digital Health Technologies | 7 months
  Participants will be asked open ended questions about their everyday experience with Digital Health Technologies. Interviews will be transcribed verbatim and analysed to identify the barriers & facilitators to Digital Health Technologies.
Strategies to enhance dignity and address barriers to Digital Health Technology adoption | 1 day
  Focus group discussions will be held with 5 participants in each group lasting around 3 hours per focus group discussion to strategise solutions to digital health technology adoption for older people.

CONTACTS AND LOCATIONS:
Overall Officials: Prof.Kathleen Galvin, PhD, Principal Investigator — University of Brighton; Dr. Theofanis Fotis, PhD, Principal Investigator — University of Brighton; Prof.Lisbeth Uhrendfeldt, PhD, Principal Investigator — Nord University
Locations (1):
- Leach Court, Brighton, East Sussex, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The investigators will follow guidelines of the European Commission on General Data Protection Regulation (GDPR), data management plan of the INNOVATEDIGNITY project and guidelines of the University of Brighton to make sure that privacy and confidentiality of the participants are retained while sharing Individual Patient Data (IPD).
Supporting Information: Study Protocol
Time Frame: Anonymised and relabelled IPD will be available at the earliest at least 1 year post publication of study results in scientific journals.
Access Criteria: Anonymised & relabelled data will be converted into metadata format by the UK Open Access Data Archive which can be accessed by other researchers for secondary analysis.
URL: http://data-archive.ac.uk

REFERENCES:
- [Background] Raleigh VS. Stalling life expectancy in the UK. BMJ. 2018 Sep 27;362:k4050. doi: 10.1136/bmj.k4050. No abstract available. PMID 30262572
- [Background] Cecula P, Behan SD, Maruthappu M. COVID-19: Challenges and opportunities in the care sector. EClinicalMedicine. 2020 May 11;23:100390. doi: 10.1016/j.eclinm.2020.100390. eCollection 2020 Jun. No abstract available. PMID 32395708
- [Background] Lawton MP. Competence, environmental press, and the adaptation of older people. In: Lawton MP, Windley PG, Byerts TO, editors. Aging and the environment: Theoretical approaches. New York: Springer. 1982.pp. 33-59.
- [Background] Wilkinson C. Evaluating the role of prior experience in inclusive design. Engineering Department. University of Cambridge.2011.
- [Background] Sleeswijk V.F., Stappers, P.J., van der Lugt, R., and Sanders, E.B.N. Contextmapping: experiences from practice. CoDesign.2005. 1 (2), 119-149. DOI: 10.1080/15710880500135987
- [Background] Hahn J. Structure of a Dissertation for a Participatory Phenomenology Design. In: Strang K.D. (eds) The Palgrave Handbook of Research Design in Business and Management. 2015.Palgrave Macmillan, New York.
- [Background] Stoecker R.Three crucial turns on the road to an adequate understanding of human dignity. In Humiliation, degradation, dehumanization. 2011; pp. 7-17. Springer, Dordrecht.
- [Background] National Institute for Health and Care Excellence. Evidence standards framework for digital health technologies.2019. https://www.nice.org.uk/Media/Default/About/what-we-do/our-programmes/evidence-standards-framework/user-guide.pdf
- [Background] University of Brighton. Brighton and Hove Digital Health Living Lab. 2018.Retrieved September 28, 2020, from https://www.brighton.ac.uk/research-and-enterprise/enterprise/enterprise-projects/brighton-and-hove-digital-health-living-lab.aspx
- [Background] United Nations. Ageing. 2019.Retrieved September 28, 2020, from https://www.un.org/en/sections/issues-depth/ageing/
- [Background] Wang S, Bolling K, Mao W, Reichstadt J, Jeste D, Kim HC, Nebeker C. Technology to Support Aging in Place: Older Adults' Perspectives. Healthcare (Basel). 2019 Apr 10;7(2):60. doi: 10.3390/healthcare7020060. PMID 30974780
- [Background] Scandurra I, Sjolinder M. Participatory Design With Seniors: Design of Future Services and Iterative Refinements of Interactive eHealth Services for Old Citizens. Med 2 0. 2013 Oct 8;2(2):e12. doi: 10.2196/med20.2729. eCollection 2013 Jul-Dec. PMID 25075235
- [Background] Renaud, K.; Karen, B.J. Judy Predicting technology acceptance and adoption by the elderly: A qualitative study. In Proceedings of the ACM International Conference Proceeding Series, Wilderness, South Africa, 6-8 October 2008; Volume 338.
- [Background] Peek ST, Wouters EJ, Luijkx KG, Vrijhoef HJ. What it Takes to Successfully Implement Technology for Aging in Place: Focus Groups With Stakeholders. J Med Internet Res. 2016 May 3;18(5):e98. doi: 10.2196/jmir.5253. PMID 27143097
- [Background] Chiu, C.-J.; Hu, Y.-H.; Lin, D.-C.; Chang, F.-Y.; Chang, C.-S.; Lai, C.-F. The attitudes, impact, and learning needs of older adults using apps on touchscreen mobile devices: Results from a pilot study. Computer Human Behaviour 2016, 63,189-197.
- [Background] Helal S, Mann W, El-Zabadani, King J, Kaddoura J, Jansen E. The gator tech smart house: a programmable pervasive space. Computer in Computer 2005;38(3):50-60.
- [Background] Sanders, E. B.-N., Generative Tools for CoDesigning in Scrivener, Ball and Woodcock, eds. Collaborative Design (London Limited: Springer-Verlag, 2000).
- [Background] Conboy-Hill, Informed Consent & Virtual Worlds, 2009. Available Online: https://www.economist.com/node/13899038
- [Background] Usher KJ, Arthur D. Process consent: a model for enhancing informed consent in mental health nursing. J Adv Nurs. 1998 Apr;27(4):692-7. doi: 10.1046/j.1365-2648.1998.00589.x. PMID 9578197
- [Background] Wherton J, Sugarhood P, Procter R, Rouncefield M, Dewsbury G, Hinder S, Greenhalgh T. Designing assisted living technologies 'in the wild': preliminary experiences with cultural probe methodology. BMC Med Res Methodol. 2012 Dec 20;12:188. doi: 10.1186/1471-2288-12-188. PMID 23256612
- [Background] Dahlberg, K., Dahlberg, H., & Nyström, M. Reflective lifeworld research (2nd ed.). 2008 Lund: Studentlitteratur.
- [Background] Personal Data Protection Commission, Guide to Basic Data Anonymisation Techniques. Singapore: 2018. Available Online: https://www.pdpc.gov.sg/-/media/Files/PDPC/PDF-Files/Other-Guides/Guide-to-Anonymisation_v1-(250118).pdf
- [Background] El Emam K. Guide to the De-Identification of Personal Health Information. CRC Press, 2013.
- [Background] European Commission (EC). Open Research Data and Data Management Plans. Brussels: ERC Scientific Council 2019. Available Online: https://erc.europa.eu/sites/default/files/document/file/ERC_info_document-Open_Research_Data_and_Data_Management_Plans.pdf
- [Background] Ramos MC. Some ethical implications of qualitative research. Res Nurs Health. 1989 Feb;12(1):57-63. doi: 10.1002/nur.4770120109. PMID 2922491